CLINICAL TRIAL: NCT06904391
Title: Building Capacity Within the NCORP Network Through an Education and Mentorship Intervention for Advanced Practice Providers (COACH-APP)
Brief Title: Education & Mentorship of Advanced Practice Providers to Increase Community-based Research Within the NCORP Network, COACH-APP Trial
Acronym: COACH-APP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00129381; NCI-2025-01059 (Other: NCI Trial Identifier)
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Other
Keywords: Mentorship, education intervention, COACH-APP
MeSH Terms: interventions — Early Intervention, Educational; Behavior Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (COACH-APP) (Experimental): APPs complete the SWOG APP Clinical Research Workshop, consisting of 6 modules, over 2 hours and receive The Advanced Practice Provider Clinical Trials Research Manual. APPs also complete 5 mentoring sessions, over 15-60 minutes each, over 12 months.
  Interventions: Other: Educational Intervention; Other: Behavioral Intervention; Other: Survey Administration; Other: Interview
- Arm II (education control) (Active Comparator): APPs receive access to the SWOG APP Clinical Research Workshop and The Advanced Practice Provider Clinical Trials Research Manual for 12 months.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Mentors (Other): The seven COACH-APP Mentors who provide the mentorship in the COACH-APP arm will also be enrolled as participants in the study.
  Interventions: Other: Survey Administration; Other: Interview
- Research Care Team Members (Other): 20 Research Care Team Members will also be enrolled in the study to participate in qualitative interviews to assess their perceptions of the COACH-APP intervention.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Educational Intervention — Receive access to SWOG APP Clinical Research workshop. Receive The Advanced Practice Provider Clinical Trials Research Manual
  Arms: Arm I (COACH-APP); Arm II (education control)
Other: Behavioral Intervention — Complete mentorship intervention
  Arms: Arm I (COACH-APP)
Other: Survey Administration — Ancillary studies
  Arms: Arm I (COACH-APP); Arm II (education control); Mentors
Other: Interview — Ancillary studies
  Arms: Arm I (COACH-APP); Mentors; Research Care Team Members

SUMMARY:
This clinical trial evaluates whether a mentorship and education intervention called COACH-APP works to improve advanced practice providers' (APPs) confidence in their ability to participate in clinical research (research self-efficacy). APPs are skilled clinicians who are routinely part of cancer care teams, but who may not routinely be part of the research care team at community oncology sites. The COACH-APP program provides focused education and structured mentorship to assist in meaningful integration to the research care team, which may increase research self-efficacy among APPs and ultimately improve patient care and access to clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare change in research self-efficacy (RSE) scores from baseline to end of study (12 months post-randomization) between APPs in the COACH-APP intervention compared to the education control.

SECONDARY OBJECTIVES:

I. To compare National Cancer Institute (NCI) Community Oncology Research Program (NCORP) engagement post-study (12-months) for APPs in the COACH-APP intervention compared to the education control.

II. To compare changes from baseline to post-study in APP ratings of research care team integration (Assessment for Collaborative Environments [ACE]-15) between the COACH-APP intervention and education control.

III. To compare practice-level NCORP and National Clinical Trial Network (NCTN) study activity as measured by total number of accruals (patient, non-patient, and organizational) and number of actively recruiting NCORP and NCTN studies over 24 months between practices with APPs receiving the COACH-APP intervention versus those in education control.

IV. Within the COACH-APP intervention group, to measure acceptability, feasibility, and appropriateness of the COACH-APP intervention for APPs and COACH-APP mentors to guide future implementation.

V. Within the COACH-APP intervention group, conduct semi-structured interviews with a sub-set of mentors, APPs, and other key research team members (collaborating oncologists and clinical research professionals) to assess:

* Va. Perceptions of feasibility, acceptability, and appropriateness of the COACH-APP intervention;
* Vb. Potential effects of the COACH-APP intervention on the research care team functioning and environment;
* Vc. Potential effects of the COACH-APP intervention on patient care quality and access to clinical trials;
* Vd. Practice-level barriers and facilitators of APP engagement in research activities.

ELIGIBILITY:
Inclusion Criteria:

* APP PRACTICE: Must have one practicing APP who can dedicate approximately 2 hours/month to participate in the intervention and study activities over a 12-month period, supported by their direct supervisor via the APP Support Statement
* APP PRACTICE: Must attest to research infrastructure that can support APP trial enrollment, as declared on the APP Practice Attestation
* APP PRACTICE: Must have submitted the APP Practice Attestation within the Study Interest Survey
* APP PRACTICE: Must have received the required APP practice ID for Oncology Patient Enrollment Network (OPEN) enrollment in the Study Selection Email prior to enrollment
* APP: Practicing nurse practitioner (NP) or physician assistant (PA) registered as an active non-physician investigators (NPIVR) within the National Cancer Institute (NCI) Registration and Credential Repository (RCR)
* APP: Treats oncology patients at practice that is actively recruiting to NCORP and/or NCTN trials
* APP: Not planning to leave their clinical position within the APP practice (defined as one or more NCORP affiliate or sub-affiliate site[s] where the APP participating in the study sees patients and clinical research activities occur) in the next 12 months at enrollment
* APP: Willing to participate in a 30-minute recorded phone interview, if selected
* APP: Completed and submitted the APP Attestation within the Study Interest Survey
* APP: Completed and submitted an APP Support Statement from their direct supervisor approving participation in this study, within the Study Interest Survey
* APP: Identify and obtain signed Research Care (RC) Team Acknowledgements from two members (defined below) of their research care team to assist them in this study. The RC team for this study will consist of an oncologist and clinical research professional (i.e., clinical research coordinator, clinical research associate clinical research nurse, etc.) that the APP collaborated with over the past 6 months or could collaborate with in the future to enroll patients on NCORP and/or NCTN trials
* APP: Must have received the required APP practice ID for OPEN enrollment in the Study Selection Email
* MENTOR: Must be a practicing APP chosen by the WF-2403 COACH-APP Study MPIs
* MENTOR: Must have the following criteria:

  * Clinical practice experience in a practice that enrolls to NCORP and/or NCTN trials.
  * Participation in a leadership role within NCTN or NCORP (i.e., serving on a Research Base committee, working group, taskforce or as a site PI)
  * Willing to complete COACH-APP mentor training.
  * Willing to complete a 30-minute recorded phone interview about their experience with the COACH-APP intervention
* RESEARCH CARE TEAM INTERVIEW: Must be an identified member of the Research Care Team for an APP assigned to the COACH-APP intervention arm. The Research Care Team will be reviewed by the APP in the 12 month survey for any changes
* RESEARCH CARE TEAM INTERVIEW: Willing to participate in a recorded phone interview (approximately 30 minutes) to assess their perceptions of the COACH-APP intervention, including feasibility, acceptability, and impact

Exclusion Criteria:

* APP PRACTICE: APP practice has an APP serving as a COACH-APP intervention mentor
* APP PRACTICE: Another APP at the same APP practice is already enrolled in this study (i.e., only 1 APP is allowed per APP practice)
* APP PRACTICE: Affiliate/sub-affiliate site(s) within this APP practice are already enrolled or are intended to be enrolled in this study under another APP practice
* APP: Has already completed the SWOG APP workshop
* APP: Served as a site principal investigator (PI) for an NCORP or NCTN study at any time
* APP: Participated as a presenter for the SWOG APP workshop
* APP: Participated on the planning committee for The Advanced Practice Provider Clinical Trials Research Manual
* APP: Participated on the planning committee for the SWOG APP workshop
* APP: Past or current member of SWOG APP Task Force Committee
* APP: Past or current member of Eastern Cooperative Oncology Group- American College of Radiology Imaging Network (ECOG-ACRIN) APP Committee
* MENTOR: Must not work at NC002-Wake Forest University Health Sciences or its affiliate/subaffiliate sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Research self-efficacy (RSE) | From baseline to 12 months post-randomization
  RSE score is calculated as sum of the 22-items measured on a 5-point Likert scale. Will be compared between the COACH-APP intervention and education control arms using a two-sample t-test.

SECONDARY OUTCOMES:
National Cancer Institute Community Oncology Research Program (NCORP) engagement | At 12 months post randomization
  Measured by the sum of 8-items measured on a 5-point Likert scale. Will be compared between the COACH-APP intervention and education control arms using linear regression.
Change in research care team integration | From baseline to 12 months post randomization
  Measured by the Assessment for Collaborative Environments (ACE)-15. Will follow the same analysis plan as for the primary outcome.
Practice-level NCORP and National Clinical Trials Network (NCTN) study activity | Up to 24 months
  Measured by total number of accruals (patient, non-patient, and organizational) and number of actively recruiting NCORP and NCTN studies. Will be compared between the COACH-APP intervention and education control arms using linear regression.
Acceptability of COACH-APP intervention (COACH-APP arm only) | At 12 months
  As measured by Acceptability of Intervention Measure (AIM). Will be summarized for the APPs in the COACH-APP intervention arm using mean and standard deviation and by capturing the percent who agree or strongly agree with the items.
Feasibility of COACH-APP intervention (COACH-APP arm only) | At 12 months
  As measured by Feasibility of Intervention Measure (FIM). Will be summarized for the APPs in the COACH-APP intervention arm using mean and standard deviation and by capturing the percent who agree or strongly agree with the items.
Appropriateness of COACH-APP intervention (COACH-APP arm only) | At 12 months
  As measured by Intervention Appropriateness Measure (IAM). Will be summarized for the APPs in the COACH-APP intervention arm using mean and standard deviation and by capturing the percent who agree or strongly agree with the items.
Perceptions of feasibility of the COACH-APP intervention | Day 1 (At time of interview)
  Measured via qualitative interview. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.
Perceptions of acceptability of the COACH-APP intervention | Day 1 (At time of interview)
  Measured via qualitative interview. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.
Perceptions of appropriateness of the COACH-APP intervention | Day 1 (At time of interview)
  Measured via qualitative interview. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.
Potential effects of the COACH-APP intervention on the research care team functioning and environment | Day 1 (At time of interview)
  Measured via qualitative interviews. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.
Potential effects of the COACH-APP intervention on patient care quality and access to clinical trials | Day 1 (At time of interview)
  Measured via qualitative interviews. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.
Practice-level barriers and facilitators of APP engagement in research activities | Day 1 (At time of interview)
  Measured via qualitative interviews. Thematic analysis of the qualitative data will be used to summarize key themes from the APP, Mentor and RC Team semi-structured interview recordings and transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (27):
- United States (27):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Illinois Cancer Care-Bloomington, Bloomington, Illinois
  - Illinois Cancer Care - Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois Cancer Care-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Cancer Care - Washington, Washington, Illinois
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maine Health Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Wake Forest NCORP Research Base, Winston-Salem, North Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu
URL: http://nctn-data-archive.nci.nih.gov/